CLINICAL TRIAL: NCT03695458
Title: Local and Systemic Effects of Photobiomodulation Therapy on Muscle Performance and Recovery Post-exercise.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Ernesto Cesar Pinto Leal Junior, Full professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 617150400
Record Dates: First submitted 2018-09-14; First posted 2018-10-04 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Phototherapy; Low-level Laser Therapy; Systemic
Keywords: phototherapy; systemic effect; recovery; performance; photobiomodulation
MeSH Terms: interventions — Phototherapy; Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Randomized, triple-blind and placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Phototherapy pad with six clusters of 12 diodes each one will be placed in both legs. Only one researcher, that will be not involved with any procedure during data collection and analysis, will know about the phototherapy program used in which leg and randomization procedure. The light aspect is the same independent of the program (active or placebo) applied and all participants will wear a opaque glasses to protect against irradiation and also assure the blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo-Control (Placebo Comparator): Photobiomodulation Therapy with the placebo program will be applied in both legs.
  Interventions: Device: Phototherapy
- irradiation effect Local (Active Comparator): Photobiomodulation Therapy with the active irradiation will be applied on the exercised leg and Photobiomodulation Therapy with the placebo program will be applied on the non-exercised leg.
  Interventions: Device: Phototherapy
- irradiation effect Systemic (Active Comparator): Photobiomodulation Therapy with the active program will be applied on non-exercised leg and Photobiomodulation Therapy with the placebo program will be applied on the exercised leg.
  Interventions: Device: Phototherapy

INTERVENTIONS:
Device: Phototherapy — The Photobiomodulation Therapy will be applied 3 minutes after MVC test in 6 points of the quadriceps muscle (2 points in vastus lateralis, 2 in rectus femoris and 2 in vastus medialis).
  Other Names: Photobiomodulation Therapy; Low-Level Laser Therapy

SUMMARY:
Recent studies with photobiomodulation therapy have shown positive results in delaying skeletal muscle fatigue and improving performance through levels of biochemical markers and variables related to exercise when this therapy was applied before exercise. Some studies suggest that photobiomodulation therapy has systemic effects, but it is not known whether therapy exerts any systemic effects on human skeletal muscle. With this factor in mind, this research aims to verify the local and systemic effects of phototherapy on muscle performance and recovery after exercise in healthy male participants. This research consists in a randomized, triple-blinded, placebo-controlled trial, with participation of 30 healthy subjects. Will be analyzed parameters related to exercise performance (peak torque in the maximum voluntary contraction test- MVC), delayed onset muscle soreness (DOMS) by visual analogue scale (VAS), and biochemical marker of muscle damage (CK) and blood Lactate (BL). The analysis will be performed before exercise protocol (baseline), after 1 minute of the exercise, and 1, 24, 48 and 72 hours after the end of exercise protocol

DETAILED DESCRIPTION:
A total of 30 healthy male non-athletes, between 18-35 years, will be randomly divided into 3 experimental groups, named "Placebo (Control)", "Local", "Systemic", according to the lower limb who will receive photobiomodulation therapy. Firstly, a blood collection will be performed by a nurse with sterile and disposable materials for posterior analysis of creatine kinase (CK) and Blood Lactate (BL). Delayed onset muscle soreness (DOMS) will be assessed with the Visual Analogue Scale (VAS) using a 10 cm line. Participants will be instructed to mark the line where their pain best fits at that time (0=no pain, 10=worst pain).Then, the maximum voluntary contraction test (MVC) will be performed, which will consist in performing 3 times of 5-sec isometric contractions of the non-dominant knee extensors in the isokinetic dynamometer device. During the execution of the MVC, the participants will be verbally encouraged to exert the greatest force at that moment. Photobiomodulation therapy will be applied 2 minutes after the MVC test in six points of non-dominant anterior thigh muscle. After irradiation, participants will perform the protocol of eccentric contractions. This protocol will be performed to induce muscle fatigue by resisting the movement of knee flexion in 5 series of 15 repetitions with 30 seconds -intervals (eccentric contractions). Assessments (blood collection, VAS and MVC) will be performed before warm-up (baseline), 1 minute after exercise protocol and 1, 24, 48 and 72 hours after eccentric exercise protocol.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals,
* Non-athletes
* Those who practice physical activity at maximal of once a week
* Between 18 and 35 years old,
* Male
* No history of musculoskeletal injury in the hip or knee previous two months of the study.
* Not be taking pharmacological agents and / or nutritional supplements, and should have frequency of 100% in all days of data collection.

Exclusion Criteria:

* Individuals who present musculoskeletal injury during the study
* Chronic joint disease in the non-dominant lower limb

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-04-14 (Actual); Study Completion 2019-05-14 (Actual)

PRIMARY OUTCOMES:
Maximum Voluntary Contraction | baseline
  An isokinetic dynamometer (System 4, Biodex®, USA) will be used to assess muscle function and also for exercise protocol. Immediately after warm-up, volunteers will perform the maximum voluntary contraction test (MVC). Volunteers will be placed on the isokinetic dynamometer seated with a 100° angle between trunk and hip, and the non-dominant leg will be positioned to 60° knee flexion (0° corresponds to the total knee extension) and attached to the seat of the dynamometer through a belt. Volunteers will also be attached to the dynamometer seat through two straps on their trunk. MVC test consists of three isometric contractions of non-dominant lower limb knee extensors with a duration of 5 seconds and 30-second intervals between contractions, the highest torque value obtained at the three contractions (peak torque) will be used for statistical analysis.
Maximum Voluntary Contraction | 1 minute after the protocol of eccentric contractions
  An isokinetic dynamometer (System 4, Biodex®, USA) will be used to assess muscle function and also for exercise protocol. Immediately after warm-up, volunteers will perform the maximum voluntary contraction test (MVC). Volunteers will be placed on the isokinetic dynamometer seated with a 100° angle between trunk and hip, and the non-dominant leg will be positioned to 60° knee flexion (0° corresponds to the total knee extension) and attached to the seat of the dynamometer through a belt. Volunteers will also be attached to the dynamometer seat through two straps on their trunk. MVC test consists of three isometric contractions of non-dominant lower limb knee extensors with a duration of 5 seconds and 30-second intervals between contractions, the highest torque value obtained at the three contractions (peak torque) will be used for statistical analysis.
Maximum Voluntary Contraction | 1 hour after the protocol of eccentric contractions
  An isokinetic dynamometer (System 4, Biodex®, USA) will be used to assess muscle function and also for exercise protocol. Immediately after warm-up, volunteers will perform the maximum voluntary contraction test (MVC). Volunteers will be placed on the isokinetic dynamometer seated with a 100° angle between trunk and hip, and the non-dominant leg will be positioned to 60° knee flexion (0° corresponds to the total knee extension) and attached to the seat of the dynamometer through a belt. Volunteers will also be attached to the dynamometer seat through two straps on their trunk. MVC test consists of three isometric contractions of non-dominant lower limb knee extensors with a duration of 5 seconds and 30-second intervals between contractions, the highest torque value obtained at the three contractions (peak torque) will be used for statistical analysis.
Maximum Voluntary Contraction | 24 hours after the protocol of eccentric contractions
  An isokinetic dynamometer (System 4, Biodex®, USA) will be used to assess muscle function and also for exercise protocol. Immediately after warm-up, volunteers will perform the maximum voluntary contraction test (MVC). Volunteers will be placed on the isokinetic dynamometer seated with a 100° angle between trunk and hip, and the non-dominant leg will be positioned to 60° knee flexion (0° corresponds to the total knee extension) and attached to the seat of the dynamometer through a belt. Volunteers will also be attached to the dynamometer seat through two straps on their trunk. MVC test consists of three isometric contractions of non-dominant lower limb knee extensors with a duration of 5 seconds and 30-second intervals between contractions, the highest torque value obtained at the three contractions (peak torque) will be used for statistical analysis.
Maximum Voluntary Contraction | 48 hours after the protocol of eccentric contractions
  An isokinetic dynamometer (System 4, Biodex®, USA) will be used to assess muscle function and also for exercise protocol. Immediately after warm-up, volunteers will perform the maximum voluntary contraction test (MVC). Volunteers will be placed on the isokinetic dynamometer seated with a 100° angle between trunk and hip, and the non-dominant leg will be positioned to 60° knee flexion (0° corresponds to the total knee extension) and attached to the seat of the dynamometer through a belt. Volunteers will also be attached to the dynamometer seat through two straps on their trunk. MVC test consists of three isometric contractions of non-dominant lower limb knee extensors with a duration of 5 seconds and 30-second intervals between contractions, the highest torque value obtained at the three contractions (peak torque) will be used for statistical analysis.
Maximum Voluntary Contraction | 72 hours after the protocol of eccentric contractions
  An isokinetic dynamometer (System 4, Biodex®, USA) will be used to assess muscle function and also for exercise protocol. Immediately after warm-up, volunteers will perform the maximum voluntary contraction test (MVC). Volunteers will be placed on the isokinetic dynamometer seated with a 100° angle between trunk and hip, and the non-dominant leg will be positioned to 60° knee flexion (0° corresponds to the total knee extension) and attached to the seat of the dynamometer through a belt. Volunteers will also be attached to the dynamometer seat through two straps on their trunk. MVC test consists of three isometric contractions of non-dominant lower limb knee extensors with a duration of 5 seconds and 30-second intervals between contractions, the highest torque value obtained at the three contractions (peak torque) will be used for statistical analysis.

SECONDARY OUTCOMES:
enzymatic activity of creatine kinase (CK) | baseline
  wil be analysis of the enzymatic activity of CK as an indirect marker of muscle damage, the initial absorbance will be read through the spectrophotometry test, use of specific reagent kits commercial manufactured (Labtest®, São Paulo - Brazil). 5 ml Blood samples, via antecubital vein puncture, will be collected in tubes by a nurse. The samples, it will be centrifuged at 3000 rpm for 20 minutes. The supernatant (serum) will then be pipetted and stored in tubes (Eppendorf ®) at -80°C for further analysis of the enzymatic activity of creatine kinase (CK).
enzymatic activity of creatine kinase (CK) | 1 minute after the protocol of eccentric contractions
  wil be analysis of the enzymatic activity of CK as an indirect marker of muscle damage, the initial absorbance will be read through the spectrophotometry test, use of specific reagent kits commercial manufactured (Labtest®, São Paulo - Brazil). 5 ml Blood samples, via antecubital vein puncture, will be collected in tubes by a nurse. The samples, it will be centrifuged at 3000 rpm for 20 minutes. The supernatant (serum) will then be pipetted and stored in tubes (Eppendorf ®) at -80°C for further analysis of the enzymatic activity of creatine kinase (CK).
enzymatic activity of creatine kinase (CK) | 1 hour after the protocol of eccentric contractions
  wil be analysis of the enzymatic activity of CK as an indirect marker of muscle damage, the initial absorbance will be read through the spectrophotometry test, use of specific reagent kits commercial manufactured (Labtest®, São Paulo - Brazil). 5 ml Blood samples, via antecubital vein puncture, will be collected in tubes by a nurse. The samples, it will be centrifuged at 3000 rpm for 20 minutes. The supernatant (serum) will then be pipetted and stored in tubes (Eppendorf ®) at -80°C for further analysis of the enzymatic activity of creatine kinase (CK).
enzymatic activity of creatine kinase (CK) | 24 hours after the protocol of eccentric contractions
  wil be analysis of the enzymatic activity of CK as an indirect marker of muscle damage, the initial absorbance will be read through the spectrophotometry test, use of specific reagent kits commercial manufactured (Labtest®, São Paulo - Brazil). 5 ml Blood samples, via antecubital vein puncture, will be collected in tubes by a nurse. The samples, it will be centrifuged at 3000 rpm for 20 minutes. The supernatant (serum) will then be pipetted and stored in tubes (Eppendorf ®) at -80°C for further analysis of the enzymatic activity of creatine kinase (CK).
enzymatic activity of creatine kinase (CK) | 48 hours after the protocol of eccentric contractions
  wil be analysis of the enzymatic activity of CK as an indirect marker of muscle damage, the initial absorbance will be read through the spectrophotometry test, use of specific reagent kits commercial manufactured (Labtest®, São Paulo - Brazil). 5 ml Blood samples, via antecubital vein puncture, will be collected in tubes by a nurse. The samples, it will be centrifuged at 3000 rpm for 20 minutes. The supernatant (serum) will then be pipetted and stored in tubes (Eppendorf ®) at -80°C for further analysis of the enzymatic activity of creatine kinase (CK).
enzymatic activity of creatine kinase (CK) | 72 hours after the protocol of eccentric contractions
  wil be analysis of the enzymatic activity of CK as an indirect marker of muscle damage, the initial absorbance will be read through the spectrophotometry test, use of specific reagent kits commercial manufactured (Labtest®, São Paulo - Brazil). 5 ml Blood samples, via antecubital vein puncture, will be collected in tubes by a nurse. The samples, it will be centrifuged at 3000 rpm for 20 minutes. The supernatant (serum) will then be pipetted and stored in tubes (Eppendorf ®) at -80°C for further analysis of the enzymatic activity of creatine kinase (CK).
Blood Lactate | baseline
  For analysis of the amount of blood lactate as an indirect marker of fatigue, a drop of blood will be collected from the first finger on the Bm-lactate strip and read through the Accutrend Plus COBAS® Monitor.
Blood Lactate | 1 minute after the protocol of eccentric contractions
  For analysis of the amount of blood lactate as an indirect marker of fatigue, a drop of blood will be collected from the first finger on the Bm-lactate strip and read through the Accutrend Plus COBAS® Monitor.
Blood Lactate | 1 hour after the protocol of eccentric contractions
  For analysis of the amount of blood lactate as an indirect marker of fatigue, a drop of blood will be collected from the first finger on the Bm-lactate strip and read through the Accutrend Plus COBAS® Monitor.
Blood Lactate | 24 hours after the protocol of eccentric contractions
  For analysis of the amount of blood lactate as an indirect marker of fatigue, a drop of blood will be collected from the first finger on the Bm-lactate strip and read through the Accutrend Plus COBAS® Monitor.
Blood Lactate | 48 hours after the protocol of eccentric contractions
  For analysis of the amount of blood lactate as an indirect marker of fatigue, a drop of blood will be collected from the first finger on the Bm-lactate strip and read through the Accutrend Plus COBAS® Monitor.
Blood Lactate | 72 hours after the protocol of eccentric contractions
  For analysis of the amount of blood lactate as an indirect marker of fatigue, a drop of blood will be collected from the first finger on the Bm-lactate strip and read through the Accutrend Plus COBAS® Monitor.
Delayed onset muscle soreness (DOMS) | baseline
  Delayed onset muscle soreness (DOMS) in the lower limb will be assessed using the Visual Analogue Pain Scale (VAS) using a 10 cm line, starting with the number 0, corresponding to no pain, and 10, corresponding to the worst possible pain. Volunteers will be instructed to mark the line where their pain best fits at that time. The evaluations will be performed prior to stretching and warm-up, 1 minute after the eccentric contractions protocol, and also 1, 24, 48, 72 hours after the protocol execution.
Delayed onset muscle soreness (DOMS) | 1 minute after the protocol of eccentric contractions
  Delayed onset muscle soreness (DOMS) in the lower limb will be assessed using the Visual Analogue Pain Scale (VAS) using a 10 cm line, starting with the number 0, corresponding to no pain, and 10, corresponding to the worst possible pain. Volunteers will be instructed to mark the line where their pain best fits at that time. The evaluations will be performed prior to stretching and warm-up, 1 minute after the eccentric contractions protocol, and also 1, 24, 48, 72 hours after the protocol execution.
Delayed onset muscle soreness (DOMS) | 1 hour after the protocol of eccentric contractions
  Delayed onset muscle soreness (DOMS) in the lower limb will be assessed using the Visual Analogue Pain Scale (VAS) using a 10 cm line, starting with the number 0, corresponding to no pain, and 10, corresponding to the worst possible pain. Volunteers will be instructed to mark the line where their pain best fits at that time. The evaluations will be performed prior to stretching and warm-up, 1 minute after the eccentric contractions protocol, and also 1, 24, 48, 72 hours after the protocol execution.
Delayed onset muscle soreness (DOMS) | 24 hours after the protocol of eccentric contractions
  Delayed onset muscle soreness (DOMS) in the lower limb will be assessed using the Visual Analogue Pain Scale (VAS) using a 10 cm line, starting with the number 0, corresponding to no pain, and 10, corresponding to the worst possible pain. Volunteers will be instructed to mark the line where their pain best fits at that time. The evaluations will be performed prior to stretching and warm-up, 1 minute after the eccentric contractions protocol, and also 1, 24, 48, 72 hours after the protocol execution.
Delayed onset muscle soreness (DOMS) | 48 hours after the protocol of eccentric contractions
  Delayed onset muscle soreness (DOMS) in the lower limb will be assessed using the Visual Analogue Pain Scale (VAS) using a 10 cm line, starting with the number 0, corresponding to no pain, and 10, corresponding to the worst possible pain. Volunteers will be instructed to mark the line where their pain best fits at that time. The evaluations will be performed prior to stretching and warm-up, 1 minute after the eccentric contractions protocol, and also 1, 24, 48, 72 hours after the protocol execution.
Delayed onset muscle soreness (DOMS) | 72 hours after the protocol of eccentric contractions
  Delayed onset muscle soreness (DOMS) in the lower limb will be assessed using the Visual Analogue Pain Scale (VAS) using a 10 cm line, starting with the number 0, corresponding to no pain, and 10, corresponding to the worst possible pain. Volunteers will be instructed to mark the line where their pain best fits at that time. The evaluations will be performed prior to stretching and warm-up, 1 minute after the eccentric contractions protocol, and also 1, 24, 48, 72 hours after the protocol execution.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline M Machado, 1, Principal Investigator — University of Nove de Julho
Locations (1):
- Universidade Nove de Julho, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vanin AA, Miranda EF, Machado CS, de Paiva PR, Albuquerque-Pontes GM, Casalechi HL, de Tarso Camillo de Carvalho P, Leal-Junior EC. What is the best moment to apply phototherapy when associated to a strength training program? A randomized, double-blinded, placebo-controlled trial : Phototherapy in association to strength training. Lasers Med Sci. 2016 Nov;31(8):1555-1564. doi: 10.1007/s10103-016-2015-7. Epub 2016 Jul 1. PMID 27371449
- [Background] Miranda EF, Vanin AA, Tomazoni SS, Grandinetti Vdos S, de Paiva PR, Machado Cdos S, Monteiro KK, Casalechi HL, de Tarso P, de Carvalho C, Leal-Junior EC. Using Pre-Exercise Photobiomodulation Therapy Combining Super-Pulsed Lasers and Light-Emitting Diodes to Improve Performance in Progressive Cardiopulmonary Exercise Tests. J Athl Train. 2016 Feb;51(2):129-35. doi: 10.4085/1062-6050-51.3.10. Epub 2016 Mar 4. PMID 26942660
- [Background] Antonialli FC, De Marchi T, Tomazoni SS, Vanin AA, dos Santos Grandinetti V, de Paiva PR, Pinto HD, Miranda EF, de Tarso Camillo de Carvalho P, Leal-Junior EC. Phototherapy in skeletal muscle performance and recovery after exercise: effect of combination of super-pulsed laser and light-emitting diodes. Lasers Med Sci. 2014 Nov;29(6):1967-76. doi: 10.1007/s10103-014-1611-7. Epub 2014 Jun 19. PMID 24942380
- [Derived] Machado CDSM, Casalechi HL, Vanin AA, de Azevedo JB, de Carvalho PTC, Leal-Junior ECP. Does photobiomodulation therapy combined to static magnetic field (PBMT-sMF) promote ergogenic effects even when the exercised muscle group is not irradiated? A randomized, triple-blind, placebo-controlled trial. BMC Sports Sci Med Rehabil. 2020 Aug 26;12:49. doi: 10.1186/s13102-020-00197-6. eCollection 2020. PMID 32864144